CLINICAL TRIAL: NCT01304615
Title: Foundations for Health: Combining Culinary Skills Training With a Lifestyle Intervention in Young Overweight Adults at Risk for Type 2 Diabetes
Brief Title: Foundations for Health
Acronym: FFH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FFH E01-1703-011
Record Dates: First submitted 2011-02-16; First posted 2011-02-25 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obese
Keywords: Overweight; Obesity; Young Adults; Energy Density; Culinary Skills; Physical Activity; Consumption of Self-made Meals; Family History of diabetes
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Web-Based (Active Comparator): Participants will receive a web-based behavioral intervention that decreases dietary energy density and increases physical activity combined with a life skills training program. Life skills training topics include stress management, coping with change, time management, and thoughts and emotions in weight control.
  Interventions: Behavioral: Decrease Energy Density of the Diet; Behavioral: Increase Steps per Day
- Web-Based plus Culinary Training (Experimental): Participants will receive a web-based behavioral intervention that decreases dietary energy density and increases physical activity combined with a hands-on culinary skills training program designed to increase food purchasing and meal self-preparation and consumption of meals low in energy density.
  Interventions: Behavioral: Decrease Energy Density of the Diet; Behavioral: Increase Steps per Day; Behavioral: Consumption of Self-made Meals

INTERVENTIONS:
Behavioral: Decrease Energy Density of the Diet — Participants will be given goals to help guide their food choices to decrease the energy density of the overall diet. The goals are to eat 10 or more foods with an ED less than 1.0 and 2 or less foods with an ED of great than 3.0 each day and to reduce portion sizes.
Behavioral: Increase Steps per Day — Participants will increase their steps per day by at least 3,000 steps per day above their baseline levels.
Behavioral: Consumption of Self-made Meals — Participants will have the goal of increasing the number of self-prepared meals that they consume to 10 or more lunch and dinner meals each week.
  Arms: Web-Based plus Culinary Training

SUMMARY:
Foundations for Health is a 12-week behavioral weight loss interventions primarily conducted via the internet aimed at helping overweight and obese young adults (ages 18-30) lose weight by increasing physical activity, decreasing the energy density of the diet, and increasing consumption of low energy dense self-made meals by providing culinary training skills.

DETAILED DESCRIPTION:
Young adulthood is recognized as a key time to focus on health promotion/disease prevention, as this time is when young individuals begin to transition to independence and thus are adopting health behaviors that will be carried into later adulthood. Unfortunately, this time period is often marked by decreases in physical activity and dietary quality. Working with young adults as they establish their first independent living situation can help set the foundation for behaviors that may aid with lifelong weight management and chronic disease prevention. Foundations for Health is the first study to examine the effect of a web-based lifestyle modification program in combination with culinary skills or lifestyle skills training sessions on weight loss, dietary intake, and meal preparation behaviors using a reduced energy dense diet in young adults with a family history of diabetes. Foundations for Health will provide a 12-week weight loss intervention for overweight and obese young adults, aged 18 to 35 years. Study participants will be randomly assigned to one of two conditions: 1) a web-based behavioral intervention that decreases dietary energy density and increases physical activity; and 2) the same intervention combined with a hands-on culinary skills training program designed to increase food purchasing and meal self-preparation and consumption of meals low in energy density. The primary aims of this feasibility study are: 1) determine if the web-based plus culinary training condition has a greater increase in food purchasing, meal preparation/cooking behaviors, and intake of self-made meals; and a greater decrease in consumption of "convenience meals" than the web-based condition at 3 months; and 2) determine if the web-based plus culinary training condition has a greater decrease in dietary energy density and percent energy from fat and a greater increase in fruit and vegetable consumption than the web-based condition at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years old.
* BMI between 25 and 45 kg/m2.
* Have type 2 diabetes or an adult family member, first or second degree relative, with type 2 diabetes.
* Have a cooking and food preparation area, along with cooking utensils, available in their current living situation.
* Consume > 3 restaurant/fast food meals/week.
* Regular and reliable internet access via a computer.

Exclusion Criteria:

* Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q).20
* Report not being able to walk for two blocks.
* Report major psychiatric diseases or organic brain syndromes.
* Are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months.
* Intend to have bariatric surgery within the time frame of the investigation.
* Intend to move outside of the metropolitan area within the time frame of the investigation.
* Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.
* Have percent body fat < 20% for females or < 13% for males.
* Live with an adult who is responsible for food purchasing and/or meal preparation.
* Have purchased a full meal plan from a college dining services program.
* Do not have regular access to transportation (needed for food purchases).
* Do not provide email contact information that is needed for access to web- based program.
* Report consuming > 10 self-made lunches or dinners per week.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Energy Density (ED) of the Diet | 3 months
  ED of the diet is will be collected using a 3 day food record and calcuated by determining the mean of the total kcals/gram weight of food consumed for each day.
Body Weight | 3 months
consumption of Self-made Meals | 3 months
  In a 3 day food record participants will report all if each meal was self-prepared, with self-prepared being defined as is a meal/food made by you that uses fruits, vegetables, low-fat sauces or herbs, lean meats, or meatless options as the main dish (entrée) of the meal. The main dish would be the component of the meal that you feel is making the largest contribution to the meal.

SECONDARY OUTCOMES:
Waist Circumference | 3 months
Steps per Day | 3 months
  Measured using the Omron HJ 720 ITC pedometer.
Percent Body fat | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hollie A. Raynor, Ph.D., Principal Investigator — University of Tennessee; Carol Costello, Ph.D., Study Chair — University of Tennessee; Ann Fairhurst, Ph.D., Study Chair — University of Tennessee
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- See also: This is the website for the Healthy Eating and Activity Laboratory (HEAL), where this program is being conducted. — http://heal.utk.edu/